CLINICAL TRIAL: NCT01338922
Title: Psychosocial Issues in Insulin Pump Therapy in Children With Type 1 DM - a Randomised Controlled Trial
Brief Title: Psychosocial Issues in Insulin Pump Therapy in Children With Type 1 Diabetes Mellitus (DM)
Acronym: pumpkin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: German Research Foundation (Other); Roche Diagnostics GmbH (Industry); University of Luebeck (Other)
Responsible Party: Principal Investigator, Verena Wagner, MD, Verena Wagner MD, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMPKIN; WA 2929/2-1/ AOBJ 582855 (Other Grant/Funding Number: German Research Foundation)
Record Dates: First submitted 2011-04-07; First posted 2011-04-20 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: open multicentre parallel randomised controlled intervention trial with waiting-list-control-group
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin pump therapy (CSII) (Experimental): Continuous subcutaneous insulin infusion therapy using different devices with marketing approval and different insulins
  Interventions: Device: Continuous subcutaneous insulin infusion therapy
- Multiple daily injection therapy (MDI) (Active Comparator): Multiple daily injection therapy using different devices with marketing approval and different insulin types
  Interventions: Device: Multiple daily injection therapy

INTERVENTIONS:
Device: Continuous subcutaneous insulin infusion therapy — Insulin is given continuously using an insulin pump. Devices are allowed having marketing approval. Insulins are permitted with marketing approval.
  Arms: Insulin pump therapy (CSII)
Device: Multiple daily injection therapy — Multiple daily injection therapy with different devices and insulin types. Devices and insulin types have to have marketing approval.
  Arms: Multiple daily injection therapy (MDI)

SUMMARY:
The effect of change in diabetes treatment from multiple daily insulin injection therapy to continuous subcutaneous insulin infusion on psychosocial outcome measures (quality of life, diabetes burden, parents stress level, fear, family conflicts) in families with children and adolescents with diabetes mellitus type 1 have been analysed. Additionally the effect on metabolic parameters (HbA1c, severe Hypoglycemia, Ketoacidosis) have been analysed.

DETAILED DESCRIPTION:
Children and adolescents currently treated with MDI and with an indication for CSII were randomized 1:1 to either starting with CSII as soon as possible or to continuing MDI while waiting six months for transmission to CSII, stratified by center. The primary outcomes were patient-reported diabetes-specific health-related quality of life , and diabetes burden of the main caregiver. We also investigated the impact of CSII on main caregiver stress, psychological well-being, fear of hypoglycemia, main caregiver's and adolescent's treatment satisfaction, family conflict, and HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 DM
* Transition to Continuous Subcutaneous Insulin Infusion (CSII)
* meeting the costs by health services
* sufficient German literacy

Exclusion Criteria:

* Remission (diabetes duration < 6 months, insulin < 0.5 i.E./kg)
* severe learning problems
* Investigator's children
* Waiting time not advised for medical reasons

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2011-04; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (HRQOL) (patient) | 6 months
  Child's HRQOL will be measured using the well-known standardized KINDL-R (KINDL) modular questionnaire. The widely used instrument provides a generic age-appropriate core-measure (24 items) and a diabetes-specific module (21 items).
Diabetes burden (main carer) | 6 months
  The main carer (parent) will report on the Overall Diabetes Burden using a one-dimensional 5-point intensity scale which was used in the pilot-study and showed sensitivity to change.
  Comment: Two primary measures are used because independent information from the child (patient) and the main carer is requested

SECONDARY OUTCOMES:
Parental stress level | 6 months
  Parental stress will be measured using the Paediatric Inventory for Parents (PIP). The 42-items instrument provides a Total Frequency Score (PIP-F), and a Total Difficulty Score (PIP-D)
Hypoglycemia fear (main carer) | 6 months
  Hypoglycemia fear will be measured using the Hypoglycaemia Fear Survey, parent version (HFS-P, Clarke et al. 1998). The 25-items instrument provides two scales: Behaviour and Worry
Family conflicts | 6 months
  Family conflict (adolescent, main carer) will be measured by the Diabetes Family Conflict Scale (DFCS). The 19 items instrument provides a DFCS Total Score
HbA1c | 6 months
  Blood samples will be collected locally with standardised equipment.The mean HbA1c value will be calculated for each patient from the last 3 measurements taken during the past six months. HbA1c values will be mathematically standardized to the Diabetes Control and Complications Trial (DCCT) -equivalent in agreement with published guidelines (Marshall& Barth 2000)
Severe Hypoglycemia International Society for Pediatric and Adolescent Diabetes (ISPAD) II/III | 6 months
  Severe hypoglycaemia grade II and grade III will be documented according to ISPAD guidelines
Diabetes treatment satisfaction | 6 months
  Treatment Satisfaction will be measured using the Diabetes Treatment Satisfaction Scale, status version (DTSQs-teen, DTSQs-parent).The validated German version will be released by MAPI (MAPI) in April 2011.

CONTACTS AND LOCATIONS:
Overall Officials: Verena Wagner, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (24):
- Germany (24):
  - Endokrinologikum Berlin, Berlin
  - Kinderklinik Charite, Berlin
  - Klinik für Kinder- und Jugendmedizin, Ruhr-Universität-Bochum, Bochum
  - Kinderkrankenhaus Kliniken der Stadt Köln GmbH, Cologne
  - PRIMA Kinderkliniken Darmstadt, Darmstadt
  - Marienhospital / Kinderklinik, Gelsenkirchen
  - Universitätsklinik Gießen, Giessen
  - Klinik am Eichert, Göppingen
  - Kinderkrankenhaus Wilhelmstift, Hamburg
  - Altonaer Kinderkrankenhaus, Hamburg
  - Gemeinschaftskrankenhaus, Herdecke
  - Praxis für Kinder- und Jugendmedizin, Herford
  - Kinderklinik Städt. Klinikum, Karlsruhe
  - UK-SH, Klinik für Allg. Pädiatrie, Kiel
  - Universität Leipzig, Kinderklinik, Leipzig
  - UK SH Campus Lübeck, Klinik für Kinder- und Jugendmedizin, Lübeck
  - Ev.Krankenhaus, Oberhausen
  - Kinderhospital Osnabrück, Osnabrück
  - Klinik f. Kinder- und Jugendmedizin, Ravensburg
  - Universitäts- Kinder- und Jugendklinik, Rostock
  - Bethlehem Gesundheitszentrum Stolberg, Stolberg
  - Olgahospital, Stuttgart
  - Universitätsklinik Tübingen, Tübingen
  - HSK-Kinderklinik, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller-Godeffroy E, Vonthein R, Ludwig-Seibold C, Heidtmann B, Boettcher C, Kramer M, Hessler N, Hilgard D, Lilienthal E, Ziegler A, Wagner VM; German Working Group for Pediatric Pump Therapy (agip). Psychosocial benefits of insulin pump therapy in children with diabetes type 1 and their families: The pumpkin multicenter randomized controlled trial. Pediatr Diabetes. 2018 Dec;19(8):1471-1480. doi: 10.1111/pedi.12777. Epub 2018 Oct 10. PMID 30302877